CLINICAL TRIAL: NCT04036890
Title: Effects of Local Minocycline Adjunctive Application in Comparison to Instrumentation Alone, in Patients With Residual Pockets Under Supportive Periodontal Therapy: a Double-blinded Randomized Controlled Clinical Trial
Brief Title: Local Minocycline in Patients Under Supportive Periodontal Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Dental Centre, Singapore (Other)
Responsible Party: Principal Investigator, Tan Wah Ching, Visiting Consultant, National Dental Centre, Singapore
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 196/2014
Record Dates: First submitted 2019-07-25; First posted 2019-07-30 (Actual); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Periodontitis
Keywords: Recurrent periodontitis; Periodontal therapy
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Intervention Model Description: Randomised, double blinded trial in parallel group
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The examiners (PI and Outcomes Assessors) will be blinded during the clinical examination of the patients. The topical antibiotic will be administered by a trained and delegated clinician who is not involved in the outcome assessment.
  Patients will be blinded to their treatment group as well.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2% minocycline hydrochloride controlled-delivery system (MHS) (Experimental): Mechanical ultrasonic/ hand instrumentation and subsequent administration of MHS on that day (Day 0) and on Day 4, at 3 months, 6 months and 9 months
  Interventions: Drug: 2% minocycline hydrochloride controlled-delivery system (MHS)
- Placebo (Placebo Comparator): Mechanical ultrasonic/ hand instrumentation and subsequent administration of a placebo gel on that day (Day 0) and on Day 4, at 3 months, 6 months and 9 months
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: 2% minocycline hydrochloride controlled-delivery system (MHS) — The test product is a highly viscous gel for local subgingival placement composing of an ointment containing micro-capsule type particles for sustained release and the active ingredient 2% minocycline gel (10mg in each syringe of 0.5g) (Periocline, SUNSTAR, Osaka, Japan). The other ingredients include magnesium chloride, hydroxyl-ethylcellulose, aminoalkylmethacrylaye copolymer, triacetin and concentrated glycerine, giving the preparation a sustained-released property. It will be applied to experimental teeth and the adjacent teeth by gently inserting the tip of a specially designed applicator until the paste flows over the gingival margin.
  Arms: 2% minocycline hydrochloride controlled-delivery system (MHS)
Drug: Placebos — It is the same gel as MHS but without active ingredient minocycline hydrochloride.
  Arms: Placebo

SUMMARY:
The aims of the present study are to assess the significance of the adjunctive effect of the subgingival application of a 2% minocycline hydrochloride controlled-delivery system (MHS) in comparison to subgingival instrumentation with application of a placebo gel, 3 months after therapy in subjects with recurrent periodontitis undergoing supportive periodontal therapy (SPT) and to assess the substantivity of the gel attributable to the adjunctive delivery of the medication that is detected at 3 months during a 9-month period of regular SPT. Recurrent periodontitis will be defined as sites with residual periodontal probing depths and bleeding on probing after completion of initial periodontal therapy. This will include both persistent and recurrent periodontitis, where persistent means the residual periodontal site after initial periodontal therapy, and recurrent means the site which was improved by initial periodontal therapy, but disease recurred.

DETAILED DESCRIPTION:
It has been reported that regular maintenance of subjects with treated periodontal disease is the key consideration in the long-term periodontal prognosis of these subjects. Periodic prophylaxis may prevent loss of clinical attachment over long periods of time even in patients with less than optimal plaque control. However, there are limitations in routine subgingival re-instrumentation especially in bleeding pockets, as only 50% of these sites improve. Furthermore, the persistence of bleeding pockets increases the risk of disease progression and tooth loss. Thus there is a need for adjuncts that may improve the outcome especially in subjects with recurrent periodontitis during SPT. Some studies reported significantly better results with subgingival administration of local minocycline in residual pockets post initial periodontal therapy over a short period of time. There are few studies assessing the efficacy of topical minocycline gel in subjects with recurrent periodontitis while in SPT, and the long term effect.

The present study will examine the significance of the adjunctive effect of the subgingival application of a 2% minocycline hydrochloride controlled-delivery system (MHS) in comparison to subgingival instrumentation with application of a placebo gel, 3 months after therapy in subjects with recurrent periodontitis undergoing supportive periodontal therapy (SPT) and to assess the substantivity of the gel attributable to the adjunctive delivery of the medication that will be detected at 3 months during a 9-month period of regular SPT.

ELIGIBILITY:
Inclusion Criteria:

* Medically healthy adults (ASA classification I-II)
* At least 21 years of age.
* Previously diagnosed with moderate to severe periodontitis and had completed at least 1 round of periodontal therapy including scaling and root-planing, oral hygiene instructions.
* Treated periodontitis patients undergoing maintenance care for at least 6 months.
* Ability to comply with 12-month study follow-up.
* Recurrent moderate to severe periodontitis with no previous systemic antibiotic therapy during initial periodontal therapy.
* At least 4 teeth present with residual PPD of ≥ 5 mm on each and a positive bleeding on probing (BOP).

Exclusion Criteria:

* Medically compromised subjects (ASA classification III-V).
* Known allergy or other severe adverse reactions to minocycline and related drugs.
* Patients who reported local and/or systemic antibiotic therapy within 3 months prior to baseline examination of the study, and were placed on antibiotics during active initial periodontal therapy.
* Patients with a plaque control record > 30%.
* Patients who had history of surgical periodontal treatment less than 5 years in the area with lesions.
* Pregnant or intend to conceive or are breast feeding.

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2016-06-03 (Actual); Primary Completion 2019-10-18 (Actual); Study Completion 2019-10-18 (Actual)

PRIMARY OUTCOMES:
Absolute change of probing pocket depth (PPD) | 3 months
  Absolute change of PPD at 3 months compared to baseline is defined as the difference between absolute patient PPD at 3 months and absolute patient PPD at baseline. For patients who have multiple trial sites, the mean of site absolute PPD will be used as their patient PPD score.

SECONDARY OUTCOMES:
Absolute change of probing pocket depth (PPD) | 6, 9,12 months
  Absolute change of PPD at 6,9 and 12 months compared to baseline are defined as the difference between absolute patient PPD at 6, 9 and 12 months and absolute patient PPD at baseline. For patients who have multiple trial sites, the mean of site absolute PPD will be used as their patient PPD score.
Percentage reduction of number of probing pocket depth (PPD) ≥ 5 mm | 3, 6, 9,12 months
  Percentage reduction of number of probing pocket depth (PPD) ≥ 5 mm at 3,6,9 and 12 months
Reduction in bleeding on probing (BOP) | 3 months vs baseline, 6 months vs baseline, 9 months vs baseline, 12 months vs baseline, 3 months vs 6 months, 3 months vs 6 months, 3 months vs 9 months, and 3 months vs 12 months.
  Defined as the difference between full mouth BOP score for each patient at two different study visits as well as the difference between bleeding score of the treatment sites at two different study visits. The comparison will be made between the following study visits: 3 months vs baseline, 6 months vs baseline, 9 months vs baseline, 12 months vs baseline, 3 months vs 6 months, 3 months vs 6 months, 3 months vs 9 months, and 3 months vs 12 months.
Change of probing attachment level (PAL) | 3, 6, 9,12 months
  Change of probing attachment level (PAL) at 3, 6, 9, 12 months compared to baseline are defined as the difference between patient PAL score at 3, 6, 9, 12 months and patient PAL score at baseline. For patients who have multiple trial sites, the mean of site PAL will be used as their patient PAL score.
Incidence of recurrent rate during experimental period. | 3, 6, 9,12 months
  The recurrent means the case of periodontal progression (attachment loss of 2mm or more) between test and groups.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-15): https://cdn.clinicaltrials.gov/large-docs/90/NCT04036890/Prot_SAP_000.pdf